CLINICAL TRIAL: NCT04723082
Title: Impacts of Sugar-Sweetened Beverage Consumption on Body Weight Regulation
Brief Title: Impacts of Sugar-Sweetened Beverage on Body Weight
Acronym: Weight
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-078-20
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Obesity
Keywords: Body fatness; Sweet taste receptors; Sugar-sweetened beverage
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We collected blood and urine samples. The researcher acknowledges the risks and ethical issues of taking biological samples, wearing correct PPE, and following the procedures for collection and handling samples. Participants will be fully aware of the study process via the PIS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The obesity epidemic is a major public health problem. Weight gain is strongly associated with an increase in the incidence of complex health conditions such as type 2 diabetes (T2D), cardiovascular disease, stroke, and cancers. Behaviours linked to food and beverage consumption can greatly affect body weight. Frequent consumption of sugar-sweetened beverages such as carbonated soft-drinks, energy and sport drinks, fruit juices from concentrate, soda and flavoured milk and water is considered to be an unhealthy dietary behaviour.

This project will investigate how variations in an individual's genes may impact their consumption of SSBs and thus body fatness. Specifically, the project will aim to investigate whether genetic variation in the taste receptors TAS1R2 and TAS1R3 can influence an individuals' perception and liking of a sweet palate and their intake of SSBs in UK. This study will be an experimental study that evaluates human body composition by different measurements. Additionally, two different biomarkers will be used for the study, such as blood and urine samples. Blood samples are the preferred source for DNA testing, rather than saliva. Urine samples will be used to look at the sugar level in the human body as a measure of body composition using deuterium dilution techniques. Around 128 adult volunteers will be recruited from Aberdeen, UK to participate in the study, which will take approximately one week to complete for each individual.

DETAILED DESCRIPTION:
To achieve this study, recruited volunteers (n=128), aged 18 years and older will visit the Rowett Institute at the University of Aberdeen on one occasion, their body composition will be measured by 3 methods: BOD POD, Tanita scales, and deuterium dilution and their consumption of SSBs will be assessed using 24h dietary recall (once in the lab and once at home over the phone). In addition, a urine sample will be collected and assessed for potential markers of sugar. Individuals will have a blood sample (up to 5 ml) taken to determine genetic variation in their taste receptors and they will also undergo a taste test using randomised tasting of a panel of 9 different sugar solutions measured in triplicate (in total they will taste 27 little cups).

The researcher will advise all the study subjects to come to a designated room in the Rowett Research Institute to complete the measurement regime at a pre-determined time between 6:30 am - 3:00 pm on their appointment day with about 2 participants per day. Each subjects measurments will take 4 hours to complete. Volunteers will complete informed consent before starting participate in the study:

Pre visit:

• Volunteers will be asked not to consume any food or drink other than water for 10 hours before their site visit, and avoid heavy exercise for 12 hours before to improve the accuracy of the body composition measurements.

Phase I:

* Volunteers will be asked to collect (fasted) urine sample to determine normal markers for sugar in their body. This will also be used to determine background isotope levels for the deuterium dilution protocol (5 minutes for collecting urine sample)
* Measurement of weight and height (BMI) (5 minutes)
* Deuterium dilution (consumption of deuterium dose; volume determined by the subjects body weight) (10 minutes).
* Demographic questionnaire (10 minutes).
* 24-h recall of SSB intake (face to face) (10 minutes). Rest Period

Phase II:

* Tanita scale (5 minutes).
* BOD POD (10 minutes). Rest Period

Phase III:

* Blood sample (15 minutes).
* Taste test (sugar solution) (50 minutes).
* Final urine sample (5 minutes).

Follow Up:

• 24-h recall SSB intake after 1 week (10 minutes).

The compulsory tests are: urine sample, measuring body composition by (deuterium, Tanita and Bod Pod), and demographic questionnaire, 24-h recall of SSB intake (face to face and phone interview), measuring weight and height (BMI) and Blood sample for genetics and the taste test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women (with no known significant health problems)
* 18 years and older (The form required me to put the maximum age, which is not stated in the protocol, so I put 100)

Exclusion Criteria:

* Less than 18 years
* Diabetic individuals
* Not living in Aberdeen city or shire
* Pregnant women
* Non-English speaker and non-able to read and understand study information sheet.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: About 128 healthy adult volunteers are required to participate in the study. They need to be living in Aberdeen City or Aberdeenshire. Participants will be requited by flyers distributing from the public who live in Aberdeen city and Aberdeenshire. Also, from the Energetics research group account on twitter.
  Participants will volunteer to take part independently.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
To establish the correlation between consumption of SSBs and body fatness. | 6 months
  Consumption of SSBs and other factors such as dietary behaviour and sociodemographic were examined previously among children and adults. Excessive consumption of SSBs in children, adolescents and adults strongly contribute to an increased risk of developing several health conditions. Statistical data that has been collected over time show the association between the consumption of SSBs and increased body weight.

SECONDARY OUTCOMES:
This research will reveal the relationship between genetic variation of taste receptors in UK adults linked with their sweet taste preferences and consumption of SSBs. | 6 months
  Genetic variation of an individual's taste receptors also plays a significant role in their preferences, and thus consumption of sugar and thus SSBs.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Hambly, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- The Rowett Institute, University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Archiving of study documents will be authorized by the sponsor at the end of the study. Essential documents will be archived for a minimum of 10 years after the completion. Documents which are not archived will be destroyed (with authorization from the sponsor). All the archived data will be stored in the HSB archive within the UoA site. Prior to archiving, during the study, material will be stored in locked filing cabinets located in the archive room in the HNU at the Rowett Institute
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: In line with MRC regulations all data will be stored for 10 years.
Access Criteria: Individual participant data (after de-identification) that underlie the results of this study will be available upon reasonable requests to investigators whose proposed used of data has been approved by an independent review committee identified for this purpose.
URL: https://www.abdn.ac.uk/achds/index.php

REFERENCES:
- See also: Genetic variation in TAS1R2 — https://pubmed.ncbi.nlm.nih.gov/20943793/
- See also: Human sweet taste, the perception and intake of sweet — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6537940/
- See also: Variation in the human TAS1R — https://pubmed.ncbi.nlm.nih.gov/16801379/
- See also: sweetened beverage consumption — https://pubmed.ncbi.nlm.nih.gov/23763695/